CLINICAL TRIAL: NCT03909906
Title: The Chronic Effects of Euphytose® on Psychological and Physiological Measures of Stress: a Randomised, Placebo-controlled, Double Blind Study in Healthy Humans
Brief Title: Chronic Effects of Euphytose® on Psychological and Physiological Measures of Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Philippa Jackson, Senior Lecturer, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 9BW1
Record Dates: First submitted 2019-04-04; First posted 2019-04-10 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Mood
Keywords: cognition; anxiety; herbal supplements
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Balanced crossover
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple masking (Participant, investigator, outcomes assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Euphytose® (Active Comparator): Euphytose® 2 tablets 3 times per day for 14 days
  Interventions: Drug: Euphytose®
- Placebo (Placebo Comparator): Matched placebo 2 tablets, 3 times per day for 14 days
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Euphytose® — (50mg Valeriana officinalis L., 40mg Passiflora incarnate L., 10mg Crataegus sp., 10mg Ballota nigra L.)
  Arms: Euphytose®
Drug: Placebo Oral Tablet — Placebo comparator
  Arms: Placebo

SUMMARY:
The aim of this study is to assess the chronic effects (14 days) of Euphytose® on psychological state, physiological stress responses and any resulting changes in gut microflora communities as compared to placebo.

DETAILED DESCRIPTION:
The aim of the proposed study is to assess the effects of chronic (14 days) supplementation with Euphytose® on psychological state with regards perceived stress and overall mood as well as psychological and physiological stress responses during a laboratory stressor. The trial will employ the Observed Multitasking Stressor (OMS), with psychological state and physiological responses assessed before and after its completion. The main mood/psychological stressor assessment will take place pre-treatment and following 14 days of treatment. Stool samples will also be collected from participants in order to assess changes in gut microflora communities at visits 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* In good physical health
* Subjects agree to abstain throughout the trial from all dietary supplements (note: protein shakes and garlic supplements are allowed)
* Body Mass Index above 18 kg/m2 and below 35 kg/m2
* Subjects are, in the opinion of the investigator, willing to participate in all scheduled visits and to adhere to all study procedures
* Subjects accept to refrain from alcohol intake 24 hours prior to Testing Visits 1-4
* Subjects do not have a current diagnosis of a significant medical condition which may interfere with the subject's ability to perform assessments and successfully completes training
* Subjects provide a personally signed and dated informed consent indicating that the subject has been informed of all pertinent aspects of the trial and understood and accepts these
* Have a bank account (required for payment)

Exclusion Criteria:

* Have any pre-existing medical condition/illness? NOTE: the exceptions to this are controlled (medicated) arthritis, asthma, high cholesterol and reflux-related conditions
* Event (personal or professional) likely to have impacted the subject's emotional and/ or psychological state within the last 8 weeks (for example but not restricted to: change of professional function/situation, death of a family member, divorce, surgery, accident, etc.)
* Event (personal or professional) likely to affect the subject's emotional, psychological or hormonal state planned during the next 8 weeks, including vaccination, important medical exam etc.
* Smoking or the use of any nicotine replacement products e.g. vaping, gum, patches (smoking within the last 3 months)
* Blood pressure >159/99 millimeters of mercury (mmHg)
* Excessive use of caffeine (> 500 mg caffeine per day) from all dietary sources
* Current intake of pharmaceuticals (excluding contraception and arthritis, cholesterol and reflux-related hormone replacement treatments (for female participants) where symptoms are stable and medications do not contraindicate the study outcomes and inhalers used as required)
* Have taken antibiotics within the last 4 weeks
* Any known active infections
* Have a recent history of (within 12 months of screening visit) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as more than 60g (men) / 40g (women) pure alcohol per day (7 / 5.5 units)
* A history of neurological or psychiatric diseases excluding anxiety or depression
* A diagnosis/treatment for a psychiatric disorder within the past 12 months (including anxiety or depression)
* A history of significant head trauma
* Have sleep disturbances and/or are taking sleep aid medication
* Have learning difficulties or dyslexia
* Have visual impairment that cannot be corrected with glasses or contact lenses (including colour blindness)
* Have frequent migraines that require medication (more than or equal to 1 per month)
* Not proficient in English equivalent to International English Language Testing System (IELTS) band 6 or above
* Are pregnant, trying to get pregnant or breast feeding
* Have any health condition that would prevent fulfillment of the study requirements
* Any condition which may interfere with the subjects ability to perform assessments
* Are employed in a job that includes night shift work
* Have no access to the internet (including via smartphone)
* Are unable to perform the computerized tests during training to the established acceptable levels for participation in this type of study.
* Have habitually used supplements, within the last month (defined as more than 3 consecutive days or 4 days in total)
* Participation in another clinical trial within 30 days prior to screening
* Any history of hypersensitivity to the investigational product or its active or inactive constituents or any food allergy or intolerance
* Non-compliant in terms of treatment consumption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Chronic treatment effects on anxiety following a psychological stressor | Following 14 days treatment
  Ratings of anxiety as defined by the Stait Trait Anxiety Inventory (STAI) - State subscale

SECONDARY OUTCOMES:
Chronic (14 days) treatment effects on general anxiety | Following 14 days treatment
  Ratings of anxiety as defined by the Stait Trait Anxiety Inventory (STAI) - Trait subscale
Chronic (14 days) treatment effects on general psychological health | Following 14 days treatment
  Ratings of general psychological health as defined by the General Health Questionnaire (GHQ-12)
Chronic (14 Days) treatment effects on stress | Following 14 days treatment
  Ratings of stress as defined by the Perceived Stress Scale (PSS) (Total score 0-40)
Chronic (14 days) treatment effects on psychological distress | Following 14 days treatment
  Ratings of stress as defined by the Profile of Mood States (POMS)
Chronic (14 days) treatment effects on subjective mood as assessed by visual analogue scales following a psychological stressor | Following 14 days treatment, measures immediately before, after and at 30, 60 and 90 minutes following a psychological stressor
  Ratings of mood (scored along a 100mm line)
Chronic (14 days) treatment effects on subjective ratings of stress as assessed by visual analogue scales following a psychological stressor | Following 14 days treatment, measures immediately before, after and at 30, 60 and 90 minutes following a psychological stressor
  Ratings of stress (scored along a 100mm line)
Chronic (14 days) treatment effects on physiological stress responses | Measures taken following 14 days treatment prior to and during a psychological stressor
  Measuring readings of galvanic skin response to determine response to psychological stressor
Chronic (14 days) treatment effects on physiological stress responses | Measures taken following 14 days treatment prior to and during a psychological stressor
  Measuring readings of heart rate response to determine response to psychological stressor
Chronic (14 days) treatment effects on other physiological stress responses | Following 14 days treatment, measures taken at baseline, immediately before, after and then at 15, 30, 60 and 90 minutes following a psychological stressor
  Measuring salivary cortisol and a-amylase to determine response to psychological stressor
Chronic (14 days) treatment effects on gut microbiota | Following 14 days treatment
  Measuring changes in gut microflora communities
Chronic (14 days) treatment effects on cognitive performance during psychological stressor | Following 14 days treatment
  Tasks include serial 3s, serial 7s, serial 17s, tracking task
7 days treatment effects on cognitive performance | Following 7 days treatment
  Tasks include simple reaction time, digit vigilance, stroop, Rapid Visual Information Processing (RVIP), peg and ball tasks
13 days treatment effects on cognitive performance | Following 13 days treatment
  Tasks include simple reaction time, digit vigilance, stroop, RVIP, peg and ball tasks
7 days treatment effects on subjective ratings of mood as assessed by visual analogue scales | Following 7 days treatment
  Ratings of mood (scored along a 100mm line)
13 days treatment effects on subjective ratings of mood as assessed by visual analogue scales | Following 13 days treatment
  Ratings of mood (scored along a 100mm line)
7 days treatment effects on subjective ratings of stress as assessed by visual analogue scales | Following 7 days treatment
  Ratings of stress (scored along a 100mm line)
13 days treatment effects on subjective ratings of stress as assessed by visual analogue scales | Following 13 days treatment
  Ratings of stress (scored along a 100mm line)
7 days treatment effects on stress | Following 7 days treatment
  Ratings of stress as defined by the Perceived Stress Scale (PSS) (Total score 0-40)
13 days treatment effects on stress | Following 13 days treatment
  Ratings of stress as defined by the Perceived Stress Scale (PSS) (Total score 0-40)
7 days treatment effects on sedation | Following 7 days treatment
  Ratings of subjective drowsiness as as defined by the Karolinska Sleepiness Scale (KSS) (Total score 1-10)
13 days treatment effects on sedation | Following 13 days treatment
  Ratings of subjective drowsiness as as defined by the Karolinska Sleepiness Scale (KSS)(Total score 1-10)

CONTACTS AND LOCATIONS:
Overall Officials: Philippa Jackson, Dr, Principal Investigator — Study Principal Investigator
Locations (1):
- Brain performance and nutrition research centre, Northumbria university, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dodd F, Kennedy D, Wightman E, Khan J, Patan M, Elcoate R, Jackson P. The chronic effects of a combination of herbal extracts (Euphytose(R)) on psychological mood state and response to a laboratory stressor: A randomised, placebo-controlled, double blind study in healthy humans. J Psychopharmacol. 2022 Nov;36(11):1243-1256. doi: 10.1177/02698811221112933. Epub 2022 Jul 23. PMID 35875924